CLINICAL TRIAL: NCT05458973
Title: Circulating Tumor DNA and BRCA Reversion Mutation in Advanced or Recurrent Ovarian Cancer Patients With Germline Mutation.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0851
Record Dates: First submitted 2022-07-05; First posted 2022-07-14 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA based on whole blood. The investigator will peripheral blood from ovarian cancer patients receiving PARP inhibitor for every three months until progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frontline cohort
- recurrent cohort

SUMMARY:
Increasing number of ovarian cancer patients are receiving PARP inhibitor as maintenance or salvage therapy. Predictive factors to PARP inhibitor other than BRCA mutation or HRD status as well as specific resistance mechanism are unknown. Thus, the objective of this study was to prospectively collect serial blood samples in ovarian cancer patients with germline BRCA mutation who receive PARP inhibitor. We investigated circulating tumor DNA (ctDNA) before patients are started on PARP inhibitor and every 3 months thereafter until progression on PARP inhibitor. Through assessment of the changes in ctDNA mutational landscape, we aimed to investigate resistance mechanism to PARP inhibitor including BRCA reversion mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of epithelial ovarian cancer,
2. Presence of germline or somatic BRCA mutation,
3. Patients receiving chemotherapy after primary debulking surgery or interval debulking surgery or patients who are planned to receive chemotherapy after recurrence on first line treatment,
4. Patients with platinum sensitive recurrence (recurrence after 6 months or longer after 1st line treatment) who are planned to receive PARP inhibitor following response to 2nd line chemotherapy.
5. Patients who recurred after 3rd or more lines of chemotherapy and are planned to receive PARP inhibitor.

Exclusion Criteria:

1. Patients who refuse to participate,
2. Patients having difficulty understanding the protocol due to language barrier

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients with germline BRCA mutation who receive PARP inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
identify resistance mechanism after PARPi | every 3 months interval until progression based on clinical surveillance (which usually ranges from 6 months to 2 years)
  Investigators will utilize baseline and post-progression samples to identify PARP resistance mechanism for each patient. For patients without baseline blood sample prior to PARP inhibitor usage, tumor Next Generation Sequencing results will be utilized. After identification of newly acquired mutations after PARP inhibitor use, these genes then will be classified into resistance mechanism category.
  Patients will undergo standard clinical surveillance, which will be based on serum CA125 and radiological assessment every 3 months interval; whole blood for ctDNA will also be collected at every 3 months interval. Upon progression based on clinical surveillance (which usually ranges from 6 months to 2 years), the corresponding whole blood-based ctDNA sample can be used as post-progression sample. The post-progression sample can then be compared with the baseline sample to inform PARP resistance mechanism.

SECONDARY OUTCOMES:
Identify pre-existing genomic profiles that may predict response to PARPi | every 3 months interval until progression based on clinical surveillance (which usually ranges from 6 months to 2 years)
  Investigators will utilize baseline blood samples to identify pre-existing genomic profiles that may predict response to PARPi. Post progression blood samples will be used to identify post-specific mechanisms that may predict response to subsequent therapy.
Identify post-progression resistance mechanisms that may predict response to subsequent therapy | every 3 months interval until progression based on clinical surveillance (which usually ranges from 6 months to 2 years)
  Investigators will utilize baseline blood samples to identify pre-existing genomic profiles that may predict response to PARPi. Post progression blood samples will be used to identify post-specific mechanisms that may predict response to subsequent therapy.
  Time frame for measurement of secondary outcome will be the same as the time frame for primary outcome. Clinical profiles such as progression-free survival with respect to PARPi, progression-free survival to post-progression subsequent therapy, and overall survival will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yun Lee, Principal Investigator — Severance hospitalYonsei University College of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YN, Shim Y, Seo J, Choi Z, Lee YJ, Shin S, Kim SW, Kim S, Choi JR, Lee JY, Lee ST. Investigation of PARP Inhibitor Resistance Based on Serially Collected Circulating Tumor DNA in Patients With BRCA-Mutated Ovarian Cancer. Clin Cancer Res. 2023 Jul 14;29(14):2725-2734. doi: 10.1158/1078-0432.CCR-22-3715. PMID 37067525